## Using Gum Arabic for Cancer Patients to Protect From Oral Mucositis Caused by Chemotherapy: An Experimental Study

NCT ID not yet assigned

15/11/2017

## Omdurman Islamic University College of Graduate Studies

Clinical Pharmacy Department

## **Informed Consent Form**

I am Abdulrazzaq Yahya Ahmed Al-Khazzan a researcher in clinical pharmacy PhD program. I will study the use of Gum Arabic for the purpose of alleviating the inflammation of the lining membrane of the mouth caused by the use of chemotherapy or radiotherapy, using Gum Arabic solution during treatment.

I would appreciate your agreement to participate in this study and you are free to participate in the study.

The information resulting from this research will be treated with complete confidentiality and will not be viewed by any person or entity other than those responsible for conducting the study, there will be no reference to your person or community in any research published on this study.

| Participant's name | Signature | Date |
|--------------------|-----------|------|